CLINICAL TRIAL: NCT03894631
Title: Intra-subject Comparison Between the Effect of Combined Phaco/Trabectome vs. Phaco/Kahook Dual Blade on Intra Ocular Pressure and Other Surgical Outcomes
Brief Title: Effect of Intra-subject Phaco/Trabectome vs. Phaco/Kahook Dual Blade on Intraocular Pressure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: State University of New York at Buffalo (Other)
Responsible Party: Principal Investigator, Asher Weiner, MD, Clinical Associate Professor, State University of New York at Buffalo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00002910
Record Dates: First submitted 2019-03-25; First posted 2019-03-28 (Actual); Last update posted 2024-07-30 (Actual); Status verified 2024-07

CONDITIONS: Glaucoma
Keywords: Kahook dual blade; Trabectome; Intraocular Pressure
MeSH Terms: conditions — Glaucoma | interventions — Phacoemulsification

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Phaco/KDB (Active Comparator): Eyes needing glaucoma and cataract extraction will receive combined KDB and phacoemulsification in one eye of a patient
  Interventions: Procedure: KDB/Phacoemulsification
- Phaco/Trabectome (Active Comparator): Contralateral eyes needing glaucoma and cataract extraction will receive combined Trabectome and phacoemulsification in contralateral eye of the same patient
  Interventions: Procedure: Trabectome/Phacoemulsification

INTERVENTIONS:
Procedure: KDB/Phacoemulsification — 50 eyes of 50 patients will receive combined KDB/phaco surgery
  Arms: Phaco/KDB
Procedure: Trabectome/Phacoemulsification — The contralateral 50 eyes of the same 50 patients will receive combined Trabectome /phaco surgery
  Arms: Phaco/Trabectome

SUMMARY:
To determine the safety and efficacy of Kahook dual blade over Trabectome in lowering intraocular pressure in glaucoma patients. Glaucoma surgery will be performed in conjunction with cataract surgery. The investigators hypothesize that the Kahook dual blade is as effective as Trabectome in lowering intra-ocular pressure (IOP), and as safe with a similar rate of post-operative complications such as hyphema.

DETAILED DESCRIPTION:
Trabectome is a type of Minimally Invasive Glaucoma Surgery (MIGS) where the Trabectome handpiece tip uses electrical current to cauterized and remove a strip of trabecular meshwork and the roof of Schlemm's canal to ease the outflow of aqueous. Kahook Dual Blade (KDB) procedure is another type of MIGS where the dual blade is used to remove the trabecular meshwork and Schlemm's canal roof to increase the aqueous outflow but without any cauterization.

Preclinical studies have evaluated the clinical outcome of Trabectome over KDB. Though Trabectome helps to lower IOP, it may remove only a portion of trabecular meshwork and possibly cause damage to surrounding tissue with leaflets of residual remaining tissue that may cause blockage of aqueous drainage. Unlike Trabectome, the KDB removes blocks of trabecular meshwork with no residual tissue leaflets, low rate of fibrosis, no damage to the surrounding tissue and lower cost. However, research studies have shown that although the Trabectome and KDB have different surgical techniques and both have surgical related risks as in any glaucoma surgery, the post-surgical clinical outcome and safety profile of Trabectome could be favorable to the KDB technique.

Few studies have evaluated the clinical outcome of Trabectome over Trabeculectomy, while few other studies evaluated Trabectome over phaco-trabectome. Some studies evaluated the clinical outcome of Trabectome alone while other studies assessed the outcome of KDB alone. Some other studies compared KDB with iStent while another study compared Trabectome versus KDB in porcine eye perfusion model. Studies have also shown that Trabectome, when combined with phaco has a higher success rate than Trabectome alone. However, due to the infancy of KDB procedure, there are no robust prospective comparison studies comparing the clinical outcome of KDB over Trabectome when combined with phacoemulsification. The aim of the study is to systematically compare the clinical outcomes of KDB over Trabectome in treating glaucoma

ELIGIBILITY:
Inclusion Criteria:

* Patients age ≥18 years old
* Patients already diagnosed with Glaucoma and Cataract in both eyes
* Patients with Primary open angle glaucoma (POAG), Low-tension glaucoma (LTG), Pseudoexfoliation glaucoma (PSXF), pigmentary glaucoma and other glaucoma types with a structurally-normal looking open angle in both eyes
* Glaucoma that is inadequately controlled on medical therapy or with the need to reduce the glaucoma medication burden
* Patients with a visually-significant cataract in both eyes
* Patients that could benefit from cataract removal combined with MIGS surgery in both eyes

Exclusion Criteria:

* Patients age less than 18 years
* Women of child bearing age
* Patients unable or unwilling to provide informed consent to participate in the study
* Aphakic and Pseudophakic patients
* Patients with primary open angle glaucoma with previously failed trabeculectomy or other glaucoma aqueous drainage surgical procedures
* Patients with a closed angle, angle neovascularization (NVG), traumatic glaucoma, or any other angle abnormality in either eye
* Patients potentially unavailable for follow up visits for the length of the study

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2019-03-06 (Actual); Primary Completion 2023-11-09 (Actual); Study Completion 2023-11-09 (Actual)

PRIMARY OUTCOMES:
Changes in intraocular pressure measurements between baseline and postoperative followup visits | 2 years
  Baseline (pre-operative condition) and post operative intraocular pressure will be measured on Day1, Week1, Months 1, 3, 6, 12, 18 and 24.

SECONDARY OUTCOMES:
Changes in visual acuity measurements measured using a Snellen Vision Chart between baseline and postoperative followup visits | 2 years
  Baseline (pre-operative condition) and post operative visual acuity will be measured on Day1, Week1, Months 1, 3, 6, 12, 18 and 24.
Changes in number of medications between baseline and postoperative followup visits | 2 years
  Baseline (pre-operative condition) and post operative number of medications list will be measured on Day1, Week1, Months 1, 3, 6, 12, 18 and 24.
Rate of post surgical complications | 2 years
  Rate of post surgical complications such as Hypotony, Corneal Edema, Hyphema, Iritis, Vitreous Hemorrhage and Cystoid Macular Edema.

CONTACTS AND LOCATIONS:
Overall Officials: Asher Weiner, MD, Principal Investigator — State University of New York at Buffalo
Locations (1):
- The Ira G. Ross Eye Institute, Buffalo, New York, United States

IPD SHARING:
Plan to Share IPD: No